CLINICAL TRIAL: NCT04061538
Title: Efficiency and Safety of Zinc Sulphate to Reduce the Duration of Acute Diarrheal Disease Between 6 and 59 Months of Age
Acronym: ESZnDiarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: UNICEF (Other)
Responsible Party: Principal Investigator, Jorge Salmeron Castro, Honorary researcher, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1474
Record Dates: First submitted 2019-08-02; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Diarrhoea;Acute; Diarrhea, Infantile
Keywords: zinc sulfate; Children; acute diarrheal diseases
MeSH Terms: conditions — Diarrhea, Infantile | interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc sulfate (Experimental): Zinc sulfate 20 mg by mouth, once a day for 10 days
  Interventions: Dietary Supplement: zinc sulfate
- Placebo (Placebo Comparator): Placebo tablet, once a day for 10 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: zinc sulfate — zinc 20mg tablets
  Arms: Zinc sulfate
Dietary Supplement: Placebo — Sugar pill manufactured to mimic zinc 20mg tablet
  Other Names: Placebo (for zinc)
  Arms: Placebo

SUMMARY:
This study evaluates the effect of zinc over the duration, severity and relapse of acute diarrheic disease, in children between 6 and 59 months of age. One study group will receive a tablet that contains 20 mg of zinc, and the other study group will receive a tablet,that does not contain zinc, it is a tablet that investigators will use as control.

DETAILED DESCRIPTION:
In Mexico acute diarrheal diseases mortality in children continues to be a public health issue, being between the main causes of morbidity and mortality, with an important load for the health systems. Consequently, there exists a necessity for the implementation of alternate strategies for this condition, nutrition being one of the pillars to strengthen.

Zinc administration during the diarrhea episode is a simple intervention for clinical picture reduction and relapse. The recommendation of including zinc in the treatment of ADD is not part of the Mexican normativity. The evaluation of the efficacy of zinc administration in Mexican children is insufficient and a program or national strategy for zinc treatment does not exist.

The objective of this study is evaluates the efficacy of oral zinc sulfate administration, during the diarrhea clinic picture in children of Mexico City.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Children attended in the sentinel centers
* Clinical diagnosis of acute diarrhea disease
* Parents have not planned moving to other location in a time period of at least one year.

Exclusion Criteria:

* Deficient intestinal absorption syndrome
* Acrodermatitis enterohepatic
* Zinc sulfate hypersensitivity
* Leucine metabolic disorders
* Secondary lactose intolerance
* Galactosemia lactase primary deficiency
* Allergy to cow milk protein
* Children that are supplemented with zinc for the last 6 months

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 529 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Diarrhea duration | 10 days
  Number of hours from the inclusion of the patient until the end of the diarrhea. The end of diarrhea was defined as the last diarrhea evacuation followed by a 48 hr period without diarrhea
Stool frequency | 10 days
  Number of stools during during the acute diarrheic disease

SECONDARY OUTCOMES:
diarrheic disease recurrence | 3 and 6 months
  Number of acute diarrheal episode, after the first episode
zinc serum concentration | 3, 9, 20, 31, 61, 91 and 121 days
  Difference of zinc serum concentration after the oral treatment for 10 days with 20 mg of zinc, and its correlation with the duration of diarrhea , the number of total stools and relapse rates

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Salmeron, PHD, Study Chair — Universidad Nacional Autonoma de Mexico; Edgar Sanchez, McS, Study Director — Universidad Nacional Autonoma de Mexico; Marcelino Esparza Aguilar, PhD, Principal Investigator — National Institute of Pediatrics in Mexico
Locations (9):
- Mexico (9):
  - Hospital Pediatrico de Coyoacan, Mexico City
  - Instituto Nacional de Pediatria, Mexico City
  - Hospital Pediatrico La Villa, Mexico City
  - Hospital Pediatrico de Iztapalapa, Mexico City
  - Hospital Pediátrico de Tacubaya, Mexico City
  - Centro de Salud Cultura Maya, Mexico City
  - Centro de Salud San Andres Totoltepec, Mexico City
  - Centro de Salud Topilejo, Mexico City
  - Hospital Materno Infantil de Xochimilco, Mexico City

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT04061538/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT04061538/Prot_SAP_001.pdf